CLINICAL TRIAL: NCT06004661
Title: An Open-label Dosimetry, Biodistribution, Tolerability and Safety Study of Lutetium (177Lu) Vipivotide Tetraxetan in Participants With Progressive PSMA-Positive Metastatic Castration-Resistant Prostate Cancer (mCRPC) With Moderately and Severely Impaired and With Normal Renal Function.
Brief Title: Study of Lutetium (177Lu) Vipivotide Tetraxetan in mCRPC Participants With Moderately and Severely Impaired and With Normal Renal Function
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAA617A12202; 2023-503925-20-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-06-29; First posted 2023-08-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Keywords: Progressive PSMA-Positive Metastatic Castration-Resistant Prostate Cancer; Prostate-specific membrane antigen; PSMA; Metastatic Castration-Resistant Prostate Cancer; mCRPC; Renal impairment; Moderately impaired renal function; Severely impaired renal function; Normal renal function; lutetium (177Lu) vipivotide tetraxetan; AAA617; Dosimetry; QTc prolongation; post marketing requirement
MeSH Terms: conditions — Renal Insufficiency | interventions — Pluvicto; gallium 68 PSMA-11

STUDY DESIGN:
Intervention Model Description: Participants confirmed for enrollment in IRT will be stratified in one of the three cohorts based on eGFR calculated (MDRD formula) at screening:
  * Cohort A: normal renal function eGFR >= 90 mL/min/1.73m2,
  * Cohort B: moderate renal impairment eGFR >= 30 to =< 59 mL/min/1.73m2
  * Cohort C: severe renal impairment eGFR >= 15 to =< 29 mL/min/1.73m2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AAA617 (Experimental): Participants will receive a dose of 7.4 GBq (200 mCi) ± 10% of AAA617 which will be administered once every 6 weeks (1 cycle) for up to 6 cycles if enrolled in Cohorts A or B. Participants with severe renal impairment (in cohort C) will receive a dose of 7.4 GBq of AAA617 for up to 3 cycles of treatment. Based on the emerging safety data and if the investigators deem the participant is still benefiting from study drug, 3 additional cycles may be administered for Cohort C participants.
  Interventions: Drug: AAA617; Drug: 68Ga-PSMA-11

INTERVENTIONS:
Drug: AAA617 — Administered intravenously once every cycles (1 cycle = 6 weeks)
  Other Names: Pluvicto; 177Lu-Lu-PSMA-617
Drug: 68Ga-PSMA-11 — Single intravenous dose of approximately 150 MBq

SUMMARY:
This study will address health authorities' requests to determine whether moderate and severe renal impairment have an impact on the biodistribution, dosimetry and safety of lutetium (177Lu) vipivotide tetraxetan (AAA617) administered to participants with progressive PSMA-positive metastatic castration-resistant prostate cancer. The study will also characterize the risk of QT prolongation of AAA617 in this participant population.

DETAILED DESCRIPTION:
This open-label, non-randomized, multicenter, single arm phase II study in mCRPC participants aims to better characterize the safety and tolerability of AAA617 in participants with moderate and severe renal impairment compared with normal renal function. Since both severe and moderate renal impairment have very low incidence within mCRPC participant population compared to participants with normal renal function, the enrollment will occur in parallel for the 3 cohorts; participants will be stratified in one of the three cohorts (A:normal, B: moderate or C: severe) based on their eGFR at screening.

All participants will undergo a 68Ga-PSMA-11 PET/CT scan at screening to confirm PSMA positivity.

Participants will receive a dose of 7.4 GBq (±10%) of AAA617 once every 6 weeks for a planned 6 cycles for cohorts A and B and 3 cycles for cohort C. Based on the emerging safety data and if the investigators deem the participant is still benefiting from study drug, 3 additional cycles may be administered for cohort C participants.

After treatment period, participants will be asked to join a long term follow up (LTFU) study to monitor their safety up to 10 years after the 1st dose of AAA617. In case of the LTFU study is not available at the time of end of treatment period (safety follow-up visit), participants will continue in Long Term Follow-up period in this study for up to one year until they can roll over into the separate LTFU study.

The primary outcome will be to determine the effect of radiation absorption in kidney and other organs at risk as well as the concentration in blood and derived PK parameters from radioactivity in blood in PSMA-positive mCRPC participants with moderate and severe renal impairment. In addition, the study will assess the relationship between drug concentrations and QTcF.

Approximately 20 participants will be enrolled in the study with at least 6 evaluable participants per cohort.

ELIGIBILITY:
Key Inclusion Criteria:

1. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
2. 68Ga-PSMA-11 Positron emission tomography (PET)/CT scan positive, and eligible as determined by the sponsor's central reader.
3. A castrate level of serum/plasma testosterone (< 50 ng/dL or < 1.7 nmol/L).
4. Documented progressive mCRPC will be based on at least 1 of the following criteria:

   * Serum/plasma Prostate-Specific Antigen (PSA) progression defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. The minimal start value is 2.0 ng/mL
   * Soft-tissue progression defined as an increase >= 20% in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of one or more new lesions.
   * Progression of bone disease: evaluable disease or new bone lesions(s) by bone scan (2+2 PCWG3 criteria)
5. Documented stable chronic renal disease without evidence of further deterioration in renal function (stable chronic renal disease is defined as no significant change in renal function within 4 weeks prior to study entry.
6. Kidney function based on eGFR by Modification of Diet in Renal Disease (MDRD) equation:

   * Normal renal function: participants with eGFR >= 90 mL/min/1.73m2
   * Moderate renal impairment: participants with eGFR >= 30 to =< 59 mL/min/1.73m2
   * Severe renal impairment: participants with eGFR >= 15 to =< 29 mL/min/1.73m2

Key Exclusion Criteria:

1. Previous treatment with PSMA-targeted radioligand therapy.
2. Previous treatment with any of the following within 6 months of enrollment confirmation: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223 or hemi-body irradiation.
3. Use of agents known to prolong the QT interval from start of screening to end of Cycle 1, unless they can be permanently discontinued for the duration of study.
4. Current severe urinary incontinence, hydronephrosis, severe voiding dysfunction, any level of urinary obstruction requiring indwelling/condom catheters. Participants with postrenal impairment, like obstructions, retroperitoneal fibrosis (eg after prostatectomy) must be excluded or first resolved to ≤ Grade 1.
5. History or current diagnosis of ECG abnormalities indicating significant risk of safety for participants participating in the study such as:

   * Concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, and clinically significant second- or third-degree AV block without a pacemaker.
   * History of familial long QT syndrome or known family history of Torsades de Pointe.
   * Resting heart rate (12 lead ECG) <60 bpm

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 20 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
Absorbed radiation dose in kidneys and selected organs | Up to 36 weeks
  The absorbed dose in kidneys and selected organs will be summarized with descriptive statistics.
Concentrations of AAA617 in blood over time | Cycle (C) 1 Day (D) 1 (pre dose, end of infusion, 20 minutes (min), 60 min, 2 and 4 hours (h) post infusion), C1 D2 (24 h post infusion), C1 D3 (48 h post infusion), C1 D4 (72 h post infusion), C1 D6 (120-144 h post infusion). Cycle=6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Blood concentration of [177Lu]Lu-PSMA-617 will be summarized with descriptive statistics.
Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of 177Lu-PSMA-617 | Cycle (C) 1 Day (D) 1 (pre dose, end of infusion, 20 minutes (min), 60 min, 2 and 4 hours (h) post infusion), C1 D2 (24 h post infusion), C1 D3 (48 h post infusion), C1 D4 (72 h post infusion), C1 D6 (120-144 h post infusion). Cycle=6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) of 177Lu-PSMA-617 | Cycle (C) 1 Day (D) 1 (2 and 4 hours (h) post infusion), C1 D2 (24 h post infusion), C1 D3 (48 h post infusion), C1 D4 (72 h post infusion), C1 D6 (120-144 h post infusion). Cycle = 6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Observed maximum plasma concentration (Cmax) of 177Lu-PSMA-617 | Cycle (C) 1 Day (D) 1 (pre dose, end of infusion, 20 minutes (min), 60 min, 2 and 4 hours (h) post infusion), C1 D2 (24 h post infusion), C1 D3 (48 h post infusion), C1 D4 (72 h post infusion), C1 D6 (120-144 h post infusion). Cycle=6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) of 177Lu-PSMA-617 | Cycle (C) 1 Day (D) 1 (pre dose, end of infusion, 20 minutes (min), 60 min, 2 and 4 hours (h) post infusion), C1 D2 (24 h post infusion), C1 D3 (48 h post infusion), C1 D4 (72 h post infusion), C1 D6 (120-144 h post infusion). Cycle=6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. The half-live will be listed and summarized using descriptive statistics
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) of 177Lu-PSMA-617 | Cycle (C) 1 Day (D) 1 (pre dose, end of infusion, 20 minutes (min), 60 min, 2 and 4 hours (h) post infusion), C1 D2 (24 h post infusion), C1 D3 (48 h post infusion), C1 D4 (72 h post infusion), C1 D6 (120-144 h post infusion). Cycle=6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-inf) will be listed and summarized using descriptive statistics.
Total systemic clearance for intravenous administration (CL) of 177Lu-PSMA-617 | Cycle (C) 1 Day (D) 1 (pre dose, end of infusion, 20 minutes (min), 60 min, 2 and 4 hours (h) post infusion), C1 D2 (24 h post infusion), C1 D3 (48 h post infusion), C1 D4 (72 h post infusion), C1 D6 (120-144 h post infusion). Cycle=6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL will be listed and summarized using descriptive statistics.
Volume of distribution during the terminal phase following intravenous elimination (Vz) of 177Lu-PSMA-617 | Cycle (C) 1 Day (D) 1 (pre dose, end of infusion, 20 minutes (min), 60 min, 2 and 4 hours (h) post infusion), C1 D2 (24 h post infusion), C1 D3 (48 h post infusion), C1 D4 (72 h post infusion), C1 D6 (120-144 h post infusion). Cycle=6 weeks
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz will be listed and summarized using descriptive statistics.
Change from baseline in eGFR | at screening and at every visit, assessed up to 1 year after last treatment
  Change from baseline of eGFR will be summarized for each post-dose (post-baseline) timepoint. The summary includes table with descriptive statistics at baseline, post-baseline time points and change from baseline to post-baseline timepoints.
Dose modifications for AAA617 | Up to 36 weeks
  Dose modifications (dose interruptions and reductions) for AAA617 will be assessed and summarized using descriptive statistics.
Dose intensity for AAA617 | Up to 36 weeks
  Dose intensity for AAA617 will be assessed and summarized using descriptive statistics.

SECONDARY OUTCOMES:
Relationship between drug concentrations and QTcF | During Cycle 1 at predose, End of Injection (EoI), 20 minutes (min), 60 min, 2 hours (h), 4h and 24h post EoI. Cycle=6 weeks
  The relationship between 177Lu-PSMA-617 plasma concentrations and ΔQTcF will be investigated using a linear mixed-effects modeling approach with ΔQTcF as the dependent variable, time-matched 177Lu-PSMA-617 plasma concentration as the explanatory variable, centered baseline QTcF (i.e., baseline QTcF for individual patient minus the population mean baseline QTcF for all patients) as an additional covariate, a fixed intercept, and a random intercept and slope per patient, when applicable (Garnett et al1).
Overall Response Rate (ORR) | From the date of 1st dose until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to approximately 36 weeks
  Objective response rate (ORR) (CR + PR) as measured by PCWG3-modified RECIST v1.1 response in soft tissue, lymph node and visceral lesions as per local review and according to PCWG3-modified RECIST v1.1. CR and PR must be confirmed by repeat assessments that should be performed not less than 4 weeks after the criteria for response are first met.
Disease Control Rate (DCR) | From the date of 1st dose until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to approximately 36 weeks
  Disease Control Rate (DCR) (CR + PR + stable disease [SD]) as measured by PCWG3-modified RECIST v1.1 response in soft tissue, lymph node and visceral lesions. DCR will be analyzed using the same analytical conventions as ORR.
PSA50 response | From screening up to 1 year
  PSA50 response is defined as the proportion of participants who have a >= 50% decrease in PSA from baseline that is confirmed by a second (the next) PSA measurement >= 4 weeks later
Potential impact of moderate and severe renal impairment on AAA617 urine PK | Cycle 1 Day 1: end of infusion to 2 hours, 2 hours to 4 hours, 4 hours to 24 hours, 24 hours to 48 hours, 48 hours to 72 hours post infusion. Cycle = 6 weeks
  Derived urine PK parameters from urine PK radioactivity data (The volume of each urine collection will be measured and the radioactivity concentration (KBq/mL) determined in order to calculate the total radioactivity excreted from the body from the start of infusion until 72h.)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Mount Sinai Hosp Med School, New York, New York, United States
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Napoli
- Spain (2):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, El Palmar, Murcia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com